CLINICAL TRIAL: NCT06760286
Title: Breathe-Easy Study: A Community-Based Trial on the Efficacy of Lung Care Solution for Improving Lung Capacity and Symptom Relief in Respiratory Conditions
Brief Title: Breathe-Easy: Food Supplement for Respiratory Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innowage Limited (Industry)
Collaborators: Mettle Networks (Unknown); Gyansanjeevani India (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: InnUK/MN/0119
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Respiration Disorders; Chronic Respiratory Conditions; Pulmonary Diseases or Conditions; Chronic Disease Management; Respiratory Tract Disorders
Keywords: Lung Care; Breathe-Easy; Dietary supplement
MeSH Terms: conditions — Respiration Disorders; Lung Diseases | interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathe-Easy (Experimental): Lung Care Solution
  Interventions: Dietary Supplement: Lung Care Solution
- Support Group (Active Comparator): Dietary advise according to the hospital routine clinical practice.
  Interventions: Other: Support treatment

INTERVENTIONS:
Dietary Supplement: Lung Care Solution — Participants in the Breathe-Easy group received the food supplement solution designed to improve lung health and respiratory function. The supplement includes natural ingredients known for their potential to reduce inflammation, improve oxygen utilization, and support overall lung capacity.
  Participants used 1 teaspoon of the supplement, prepared as a tea decoction, twice daily.
  Other Names: Bionutriva
  Arms: Breathe-Easy
Other: Support treatment — Participants in this group engaged in guided lifestyle modifications aimed at improving respiratory health. This included dietary recommendations as part of clinical practice.
  Arms: Support Group

SUMMARY:
The trial aims to assess the effectiveness of a natural lung care solution and a food supplement in improving lung function, capacity, and alleviating symptoms associated with respiratory conditions like asthma, COPD, and chronic bronchitis.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and older.
* Diagnosed with a chronic respiratory condition (e.g., asthma, COPD).
* No known allergies to ingredients in the supplement.
* Ability to provide informed consent and comply with study procedures.

Exclusion Criteria:

* Acute respiratory infection within the last 30 days.
* Current participation in another clinical trial.
* History of severe adverse reactions to similar supplements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2024-05-12 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Changes in pulmonary function | Change in forced expiratory volume (FEV1) from baseline to 12 weeks.
  Differences in forced expiratory volume measured by spirometry

SECONDARY OUTCOMES:
Symptom Severity Scores | Change in symptom scores from baseline to 12 weeks.
  Symptom severity assessed to measure the impact of the interventions on respiratory symptoms such as shortness of breath, coughing, wheezing, and chest tightness.
Quality of Life (QoL) | Change in quality of life from baseline to 12 weeks.
  QoL measured using the St. George's Respiratory Questionnaire (SGRQ)

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Shinde, Study Chair — Mettle Networks, UK; Dr Neha Sharma, Study Director — Innowage UK; Dr Bidyanand Jha, Study Director — Lexicon MILE, India; Dr Sadhana Sharma, Principal Investigator — Gyansanjeevani India; Dr Mridu Sharma, Study Chair — Mettle Networks, UK; Dr. Pradyuman S Rathore, Principal Investigator — Lexicon MILE, India
Locations (1):
- Gyansanjeevani India, Jaipur, India

IPD SHARING:
Plan to Share IPD: Undecided